CLINICAL TRIAL: NCT07039422
Title: Exploratory Study of Ianalumab in Adults With Primary Immune Thrombocytopenia (ITP) and Warm-antibody Autoimmune Hemolytic Anemia (wAIHA) Who Have Previously Benefited From Ianalumab (VAY RE-HIT)
Brief Title: Study of Ianalumab in Adults With Primary Immune Thrombocytopenia (ITP) and Warm-antibody Autoimmune Hemolytic Anemia (wAIHA) Who Have Previously Benefited From Ianalumab
Acronym: VAY RE-HIT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVAY736Q12202B; 2024-518231-11-00 (Other: EU CTIS)
Expanded Access: NCT07244289 (Available)
Record Dates: First submitted 2025-05-05; First posted 2025-06-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Primary Immune Thrombocytopenia; Warm Autoimmune Hemolytic Anemia
Keywords: Primary Immune Thrombocytopenia (ITP); ITP; Warm Autoimmune Hemolytic Anemia (wAIHA); wAIHA; VAY736; Ianalumab; B-cell depletion; B-cell Activating Factor Receptor (BAFF-R) blockade
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — ianalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded will be maintained at least until parent studies are unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment arm 1 (Experimental): Participants will receive ianalumab lower dose
  Interventions: Biological: Ianalumab
- Treatment arm 2 (Experimental): Participants will receive ianalumab higher dose
  Interventions: Biological: Ianalumab

INTERVENTIONS:
Biological: Ianalumab — Concentrate for solution for infusion for intravenous use
  Other Names: VAY736

SUMMARY:
This study is intended to explore the efficacy and safety of a second course of ianalumab after experiencing treatment failure in the pivotal Primary Immune Thrombocytopenia (ITP) trials (CVAY736I12301, CVAY736Q12301) and after loss of durable response in the pivotal Warm Autoimmune Hemolytic Anemia (wAIHA) trial (CVAY736O12301).

DETAILED DESCRIPTION:
This is a multicenter, Phase 2 exploratory study to assess the efficacy and safety of a second course of ianalumab in adults with ITP and wAIHA who have previously benefited from ianalumab.

All participants will receive ianalumab at the dose of study treatment from which they previously derived benefit.

After completion of the screening period, participants who do not meet treatment failure criteria during treatment period will enter the safety and efficacy follow-up, whereas participants who reported a treatment failure during the treatment period will enter the safety follow-up only.

The study will end once all participants have completed safety and/or efficacy follow-up since their last dose of ianalumab or discontinued the study earlier.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained prior to participation in the study.
* Male or female participants aged 18 years and older on the day of signing informed consent

Primary ITP patients:

* Previously enrolled and treated either with ianalumab/placebo in addition to first-line corticosteroids on protocol CVAY736I12301 or with ianalumab/placebo in addition to eltrombopag in the second line on protocol CVAY736Q12301, and who experienced treatment failure (TF) by parent trial definition ≥ 2 years after the last infusion of ianalumab/placebo
* Rescue medication and/or bridging therapy are allowed to be started within the 28 days prior to screening; platelet count results obtained prior to the start of the therapy must be used to assess eligibility and have to be collected within 30 days prior to screening

For Primary or secondary wAIHA patients:

* Previously documented by a positive direct antiglobulin test (DAT) specific for anti-IgG or anti-IgA, previously enrolled and treated with ianalumab/placebo in blinded cohort or placebo followed by crossover to open label ianalumab in protocol CVAY736O12301, having experienced durable response lasting beyond 2 years from the last infusion of ianalumab/placebo in blinded cohorts or a durable response beyond week 20 from last dose of first course of ianalumab in the crossover arm.
* Relapsed wAIHA with hemoglobin concentration ≥5 g/dL and <10 g/dL and presence of symptoms related to anemia during screening or within 14 days before screening window or within 28 days before screening window if rescue medication/bridging therapy has been initiated.
* Rescue medication and/or bridging therapy are allowed to be started during the screening and within 28 days prior to screening; hemoglobin level result for eligibility assessment needs to be obtained prior to the start of the treatment within 30 days prior to screening
* Supportive care is allowed in the case the participant received it in the parent trial when the relapse occurred and has remained stable at least 4 weeks prior screening

Exclusion Criteria:

* Evans syndrome or any cytopenia other than thrombocytopenia (for ITP participants) or anemia (for wAIHA), except for grade 1 anemia due to blood loss or iron deficiency.
* Secondary wAIHA with BM involvement for wAIHA patients
* Current life-threatening bleeding or history of life-threatening bleeding due to thrombocytopenia
* Therapy for ITP or wAIHA other than ianalumab/placebo, bridging/rescue therapies and supportive care prior to the beginning of the screening window
* After primary analysis of each respective parent trial, participants whose treatment was unblinded and who received placebo only will be excluded.
* ITP participants only: Participants with concurrent coagulation disorders and/or receiving anti-platelet or anti-coagulant medication except for low dose of acetylsalicylic acid (≤150 mg per day)

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2030-08-30 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
Treatment failure free (yes, no) for participants with Immune Thrombocytopenia (ITP) | From treatment start date until the events indicative of treatment failure (up to 2 years after last dose)
  Treatment failure free (yes, no) by 12 months after start of second course of ianalumab at assigned dose.
Durable response for participants with Warm Autoimmune Hemolytic Anemia (wAIHA) | At least 8 consecutive weeks, between week 9 and week 25
  Durable response (hemoglobin (Hb) ≥ 10 g/dL and ≥ 2 g/dL increase from baseline) for a period of at least 8 consecutive weeks, between W9 and W25 in the absence of rescue or prohibited treatment prior to that durable response achievement.

SECONDARY OUTCOMES:
Response rate in participants with ITP only | from treatment start to end of study (up to 2 years after last dose)
  Percentage of participants with ITP achieving a response among all participants who received a second course of ianalumab, and among cohorts and/or group of cohorts.
Complete response rate in participants with ITP only | from treatment start to end of study (up to 2 years after last dose)
  Percentage of participants with ITP achieving a complete response among all participants who received a second course of ianalumab, and among cohorts and/or group of cohorts.
Number and percentage of participants receiving new ITP therapy only | from treatment start to end of study (up to 2 years after last dose)
  Number and percentage of participants who need new ITP therapy among all the participants who received a second course of ianalumab, and among cohorts and/or group of cohorts.
Response and complete response in participants with wAIHA only | from treatment start to end of study (up to 2 years after last dose)
  Percentage of participants with wAIHA achieving a response and complete response among all participants who received a second course of ianalumab and among cohorts and/or group of cohorts.
Number and percentage of participants receiving new wAIHA therapy only | from treatment start to end of study (up to 2 years after last dose)
  Number and percentage of participants who need new wAIHA therapy among all the participants who received a second course of ianalumab, and among cohorts and/or group of cohorts.
Number and percentage of participants receiving rescue treatment | from treatment start to end of study (up to 2 years after last dose)
  Number and percentage of participants who need rescue treatment among all the participants who received a second course of ianalumab, and among cohorts and/or group of cohorts.
Number of severe infections and percentage of participants with severe infection | from treatment start to end of study (up to 2 years after last dose)
  This is to assess the safety profile of ianalumab.
Ianalumab concentration in serum | after first dose (pre dose 0 and 672 hours) and at study end (up to 2 years after last dose of Ianalumab)
  Assess the pharmacokinetics of a second course of ianalumab treatment.
Incidence of anti-ianalumab antibodies in serum (ADA assay) over time | up to end of treatment (Week 16), end of study (up to 2 years after last dose of Ianalumab)
  Anti-drug antibodies (ADA) will be evaluated in samples collected from all participants to assess the immunogenicity of Ianalumab.
Titer of anti-ianalumab antibodies in serum (ADA assay) over time | up to end of treatment (Week 16), end of study (up to 2 years after last dose of Ianalumab)
  Assess the immunogenicity of second course of ianalumab treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Ostrava, Poruba, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com